CLINICAL TRIAL: NCT04652102
Title: COVID-19: A Phase 2b/3, Randomized, Observer-Blinded, Placebo-Controlled, Multicenter Clinical Study Evaluating the Efficacy and Safety of Investigational SARS-CoV-2 mRNA Vaccine CVnCoV in Adults 18 Years of Age and Older
Brief Title: A Phase 2b/3, Randomized, Observer-Blinded, Placebo-Controlled, Multicenter Clinical Study Evaluating the Efficacy and Safety of Investigational SARS-CoV-2 mRNA Vaccine CVnCoV in Adults 18 Years of Age and Older
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CV-NCOV-004; 2020-003998-22 (EudraCT Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-03 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2023-11

CONDITIONS: Covid19; SARS-CoV-2
Keywords: Vaccine
MeSH Terms: conditions — COVID-19 | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The randomized observer-blinded phases of this study are participant and investigator blinded. This is followed by an open-label phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Randomized Observer-blinded Phase 2b: CVnCoV vaccine (Experimental): Participants will be vaccinated with CVnCoV 12 µg vaccine on Day 1 and Day 29 in the deltoid area, preferably in the non-dominant arm.
  Interventions: Biological: CVnCoV
- Randomized Observer-blinded Phase 2b: Placebo (Placebo Comparator): Participants will be administered the matching placebo on Day 1 and Day 29 in the deltoid area, preferably in the non-dominant arm.
  Interventions: Biological: Placebo
- Randomized Observer-blinded Phase 3: CVnCoV vaccine (Experimental): Participants will be vaccinated with CVnCoV 12 µg vaccine on Day 1 and Day 29 in the deltoid area, preferably in the non-dominant arm.
  Interventions: Biological: CVnCoV
- Randomized Observer-blinded Phase 3: Placebo (Placebo Comparator): Participants will be administered the matching placebo on Day 1 and Day 29 in the deltoid area, preferably in the non-dominant arm.
  Interventions: Biological: Placebo
- Open-label Phase (Experimental): After unblinding, the trial will shift from a randomized observer-blinded to an open-label design, and the following cohorts will be defined:
  Cohort A: participants who received at least 1 dose of CVnCoV in the randomized observer-blinded phases and choose to receive an authorized/licensed vaccine for preventing COVID-19 (AV) as standard of care through their national vaccination program.
  Cohort B: participants who received at least 1 dose of CVnCoV in the randomized observer-blinded phases and choose to remain in the trial without receiving any AV.
  Participants on the placebo arm will be withdrawn.
  Interventions: Biological: Authorized/licensed vaccines for preventing COVID-19 (AV) as standard of care through their national vaccination program

INTERVENTIONS:
Biological: CVnCoV — Intramuscular (IM) injection.
  Other Names: CV07050101
  Arms: Randomized Observer-blinded Phase 2b: CVnCoV vaccine; Randomized Observer-blinded Phase 3: CVnCoV vaccine
Biological: Placebo — Intramuscular (IM) injection.
  Arms: Randomized Observer-blinded Phase 2b: Placebo; Randomized Observer-blinded Phase 3: Placebo
Biological: Authorized/licensed vaccines for preventing COVID-19 (AV) as standard of care through their national vaccination program — Intramuscular (IM) injection will be received as standard of care (SoC) outside the study.
  Arms: Open-label Phase

SUMMARY:
The primary objective of the randomized observer-blinded phase 2b/3 part of this trial is to demonstrate the efficacy of a 2-dose schedule of CVnCoV in the prevention of first episodes of virologically-confirmed cases of COVID-19 of any severity in SARS-CoV-2 naïve participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 years of age or older.
* Be willing and able to provide written informed consent prior to initiation of any trial procedures.
* Expected compliance with protocol procedures and availability for clinical follow-up through the last planned visit.
* Females of non-childbearing potential defined as follows: surgically sterile (history of bilateral tubal ligation/occlusion, bilateral oophorectomy or hysterectomy) or postmenopausal {defined as amenorrhea for ≥12 consecutive months prior to screening (Day 1) without an alternative medical cause}. A follicle-stimulating hormone (FSH) level may be measured at the discretion of the Investigator to confirm postmenopausal status.
* Females of childbearing potential: negative pregnancy test (human chorionic gonadotropin [hCG]) within 24 hours prior to each trial vaccination on Day 1 and Day 29.
* Females of childbearing potential must use highly effective methods of birth control from 2 weeks before the first administration of the trial vaccine until 3 months following the last administration. The following methods of birth control are considered highly effective when used consistently and correctly:

  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal);
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable);
  * Intrauterine devices;
  * Intrauterine hormone-releasing systems;
  * Bilateral tubal ligation;
  * Vasectomized or infertile partner;
  * Sexual abstinence {periodic abstinence (e.g., calendar, ovulation, symptothermal and post-ovulation methods) and withdrawal are not acceptable}.

Exclusion Criteria:

* History of virologically-confirmed COVID-19 illness.
* For females: pregnancy or lactation.
* Use of any investigational or non-registered product (vaccine or drug) within 28 days preceding the administration of trial vaccine or planned use during the trial.
* Receipt of any licensed vaccines within 28 days (for live vaccines) or 14 days (for inactivated or any other vaccines) prior to administration of the first trial vaccine.
* Prior administration of any investigational SARS-CoV-2 vaccine or another coronavirus (SARS-CoV, Middle East Respiratory Syndrome-CoV) vaccine or planned used during the trial.
* Any treatment with immunosuppressants or other immune-modifying drugs (including but not limited to anabolic steroids, corticosteroids, biologicals and methotrexate) for > 14 days total within 6 months preceding the administration of trial vaccine or planned use during the trial. For corticosteroid use, this means prednisone or equivalent, 0.5 mg/kg/day for 14 days or more. The use of inhaled, topical, or localized injections of corticosteroids (e.g., for joint pain/inflammation) is permitted.
* Any medically diagnosed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination including known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV); current diagnosis of or treatment for cancer including leukemia, lymphoma, Hodgkin disease, multiple myeloma or generalized malignancy; chronic renal failure or nephrotic syndrome; and receipt of an organ or bone marrow transplant.
* History of angioedema (hereditary or idiopathic) or history of any anaphylactic reaction.
* History of potential immune-mediated disease (pIMD).
* History of allergy to any component of CVnCoV.
* Administration of immunoglobulins or any blood products within 3 months prior to the administration of trial vaccine or planned receipt during the trial.
* Participants with a significant acute or chronic medical or psychiatric illness that, in the opinion of the Investigator, precludes trial participation (e.g., may increase the risk of trial participation, render the participant unable to meet the requirements of the trial, or may interfere with the participant's trial evaluations). These include severe and/or uncontrolled cardiovascular disease, gastrointestinal disease, liver disease, renal disease, respiratory disease, endocrine disorder, and neurological and psychiatric illnesses. However, those with controlled and stable cases can be included in the trial.
* Participants with impaired coagulation or any bleeding disorder in whom an IM injection or a blood draw is contraindicated.
* Foreseeable non-compliance with the trial procedure as judged by the Investigator.

Roll-over Criteria for the Open-label Phase:

* Participants must have received at least 1 dose of CVnCoV during the randomized observer blinded phase.
* Participants must provide additional written informed consent to be eligible for the open label phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39680 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- Argentina (9):
  - Instituto de Investigaciones Clinicas Quilmes, Buenos Aires
  - Hospital Interzonal General Agudos Prof. Dr. Ramon Carrillo, Buenos Aires
  - Hospital Interzonal General de Agudos Vicente Lopez y Planes, Buenos Aires
  - Hospital Zonal General de Agudos Descentralizado Evita Pueblo de Berazategui, Buenos Aires
  - Fundación Cenit Para La Investigación En Neurociencias, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata
  - Sanatorio Parque, Rosario
  - Corporación Médica Sanatorio, San Martín
  - Instituto De Investigaciones Clinica Zarate, Zárate
- Belgium (3):
  - Cohezio - Bruxelles, Brussels
  - Mensura, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Colombia (3):
  - Clínica de la Costa, Barranquilla
  - CAIMED - Bogota Clinical Research Center, Bogotá
  - Centro de Estudios en Infectología Pediátrica (CEIP), Cali
- Dominican Republic (4):
  - Fundacion Dominicana de Perinatologia Pro Bebe, Santo Domingo
  - Instituto Dermatológico Dominicano y Cirugía de Piel Dr. Huberto Bogaert Díaz, Santo Domingo
  - Clínica Cruz Jiminian, Santo Domingo
  - Hospital General Regional Marcelino Vélez Santana, Santo Domingo
- Germany (3):
  - Uniklinik Köln, Cologne
  - Ludwig-Maximilians-Universität München, München
  - Universitätsklinikum Tübingen - Institut für Tropenmedizin, Reisemedizin und Humanparasitologie, Tübingen
- Mexico (6):
  - Panamerican Clinical research Mexico (Guadalajara), Guadalajara
  - Panamerican Clinical Research Mexico S.A. DE C.V., Juriquilla
  - Instituto Nacional De Ciencias Medicas Y Nutricion Salvador Zubiran, Mexico City
  - CAIMED - México, Mexico City
  - Unidad de Medicina Especializada SMA, San Juan del Río
  - Centro Medico Zambrano Hellion TecSalud, San Pedro Garza García
- Netherlands (3):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Amsterdam Universitair Medische Centra - Academisch Medisch Centrum, Amsterdam
  - The Julius Center - Utrecht Science Park - Stratenum, Utrecht
- Panama (4):
  - Centro De Vacunacion Internacional - CEVAXIN Chorreras, Panama City
  - Instituto de Investigaciones Científicas y Servicios de Alta Tecnología, Panama City
  - Centro De Vacunacion Internacional - CEVAXIN 24 Diciembre, Panama City
  - Centro de Vacunacion Internacional - CEVAXIN Avenida Mexico, Panama City
- Peru (8):
  - Centro de Investigaciones Tecnológicas, Biomédicas y Medioambientales, Callao
  - Hospital de Chancay y Servicios básicos de Salud, Chancay
  - Clinica Medica San Martin, Ica
  - Instituto de Investigación Nutricional - Las Gardenias, Lima
  - Instituto de Investigación Nutricional - San Carlos, Lima
  - Instituto de Investigación Nutricional, Lima
  - Asociación Civil Impacta Salud y Educación, Lima
  - Centro de Investigación para ensayos Clínicos UPCH, Lima
- Spain (3):
  - OSI Eskerraldea-Enkarterri-Cruces/Hospital Universitario Cruces, Barakaldo
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Clínico San Carlos, Madrid

REFERENCES:
- [Derived] Kremsner PG, Ahuad Guerrero RA, Arana-Arri E, Aroca Martinez GJ, Bonten M, Chandler R, Corral G, De Block EJL, Ecker L, Gabor JJ, Garcia Lopez CA, Gonzales L, Granados Gonzalez MA, Gorini N, Grobusch MP, Hrabar AD, Junker H, Kimura A, Lanata CF, Lehmann C, Leroux-Roels I, Mann P, Martinez-Resendez MF, Ochoa TJ, Poy CA, Reyes Fentanes MJ, Rivera Mejia LM, Ruiz Herrera VV, Saez-Llorens X, Schonborn-Kellenberger O, Schunk M, Sierra Garcia A, Vergara I, Verstraeten T, Vico M, Oostvogels L; HERALD Study Group. Efficacy and safety of the CVnCoV SARS-CoV-2 mRNA vaccine candidate in ten countries in Europe and Latin America (HERALD): a randomised, observer-blinded, placebo-controlled, phase 2b/3 trial. Lancet Infect Dis. 2022 Mar;22(3):329-340. doi: 10.1016/S1473-3099(21)00677-0. Epub 2021 Nov 23. PMID 34826381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was performed in Argentina, Belgium, Colombia, the Dominican Republic, Germany, Mexico, the Netherlands, Panama, Peru and Spain between 11 December 2020 and 10 June 2022.
Pre-assignment Details: Of the 39680 participants who were randomized, 39540 participants received at least one dose vaccine.
Groups:
- CVnCoV 12 μg Vaccine: Participants in the Phase 2b and Phase 3 periods were vaccinated with CVnCoV 12 μg as an intramuscular injection by needle in the deltoid area, preferably in the non-dominant arm, on Day 1 and Day 29.
- Placebo: Participants in the Phase 2b and Phase 3 periods were vaccinated with matching placebo as an intramuscular injection by needle in the deltoid area, preferably in the non-dominant arm, on Day 1 and Day 29.
Period: Overall Study
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Started | 19787 | 19753
Phase 2b Participants | 2007 | 1987
Phase 3 Participants | 17780 | 17766
Rolled Over to Open-Label Phase | 8513 | 0
Completed | 11451 | 4161
Not Completed | 8336 | 15592
Not completed — Adverse Event | 14 | 13
Not completed — Subject Received Alternative Authorised Vaccine | 1407 | 6552
Not completed — Physician Decision | 78 | 40
Not completed — Study Ended by Sponsor | 64 | 17
Not completed — Withdrawal by Subject | 4625 | 5594
Not completed — Lost to Follow-up | 2019 | 1082
Not completed — Protocol Specified Withdrawal Criterion Met | 49 | 2230
Not completed — Miscellaneous | 80 | 64

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: Included all participants randomized into Phase 2b or 3 who received at least one dose of CVnCoV or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | CVnCoV 12 μg Vaccine | Placebo | Total
Number analyzed (Participants) | 19787 | 19753 | 39540
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (14.49) | 43.0 (14.50) | 43.0 (14.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8935 | 8936 | 17871
  Male | 10852 | 10817 | 21669
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14732 | 14740 | 29472
  Not Hispanic or Latino | 4960 | 4932 | 9892
  Unknown or Not Reported | 95 | 81 | 176
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 9012 | 8989 | 18001
  Race: Black or African American | 383 | 356 | 739
  Race: Asian Indian | 18 | 10 | 28
  Race: Chinese | 21 | 22 | 43
  Race: Filipino | 1 | 3 | 4
  Race: Japanese | 5 | 0 | 5
  Race: Korean | 0 | 2 | 2
  Race: Vietnamese | 9 | 9 | 18
  Race: American Indian or Alaska Native | 2492 | 2485 | 4977
  Race: Other | 7797 | 7812 | 15609
  Race: Not Reported | 34 | 44 | 78
  Race: Unknown | 15 | 21 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a First Episode of Virologically-confirmed {Reverse Transcription Polymerase Chain Reaction (RT-PCR) Positive} Case of COVID-19 of Any Severity
Description: A case of COVID-19 meeting the definition for primary efficacy analysis was defined as follows:
  * Virologically-confirmed case of COVID-19 (of any severity) defined as a positive SARS-CoV-2 specific RT-PCR test in a person with clinically symptomatic COVID-19.
  * Symptom onset ≥ 15 days after second trial vaccination.
  * First episode of virologically-confirmed COVID-19, i.e. the participant must not have had a history of virologically-confirmed COVID-19 illness at enrollment or have had developed a case of virologically-confirmed COVID-19 before 15 days after the second trial vaccination.
  * Participant was SARS-CoV-2 naïve at baseline and Day 43 (defined as seronegative to N protein in the blood samples collected at baseline and Day 43).
  * Primary efficacy cases were confirmed by an Adjudication Committee.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Day 44 to Day 393
Population: Efficacy Analysis Set (EAS): All participants randomized in Phase 2b or Phase 3 who received both doses of trial vaccine, had not developed a virologically-confirmed case of COVID-19 before trial entry or before 15 days after the second vaccination & were SARS-CoV-2 naïve at baseline & Day 43. Participants must have not developed an asymptomatic case of SARS-CoV-2, not stopped the trial, not received an AV for preventing COVID-19 or been unblinded prior to 15 days after the second vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 12851 | 12211
Participants | 83 | 145
Statistical Analysis 1: Comparison: CVnCoV 12 μg Vaccine vs Placebo; Proportion of cases coming from the CVnCoV group among all cases; Test type: Superiority; Proportion = 0.364, 95.826% CI 2-sided [0.299 to 0.433] — Derived from an exact 2-sided 95.826% Pearson-Clopper confidence interval (CI) on proportion of cases coming from the CVnCoV group among all cases
Statistical Analysis 2: Comparison: CVnCoV 12 μg Vaccine vs Placebo; Vaccine efficacy (VE) calculated as VE = 1 - p/(1-p) *1/r where p represents the proportion of cases coming from the CVnCoV group among all cases and r represents the ratio of total follow-up time of subjects in the CVnCoV group over the total follow-up time of subjects in the placebo group; Test type: Other; p = 0.01600, Exact Binomial Test — 1-sided p-value from the exact binomial test on proportion of cases coming from the CVnCoV group among all cases (equivalent to a test on VE with H0: VE ≤30%). Statistically significant if lower than 0.02087; Vaccine Efficacy = 48.2, 95.826% CI 2-sided [31.0 to 61.4] — 2-sided 95.826% CI on VE, derived from the exact 2-sided 95.826% Pearson-Clopper CI on proportion of cases coming from the CVnCoV group among all cases

2. Primary Outcome: Number of Participants Who Experienced One or More Medically-attended Adverse Events (AE)
Description: Medically-attended AEs were defined as AEs with medically-attended visits that were not routine visits for physical examination or vaccination, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Clinic visits for COVID-19 testing resulting in negative test results were not considered as medically attended visits, if there is no confirmed diagnosis and no prescribed concomitant medication.
  The Investigator assessed the relationship between trial vaccine and occurrence of each AE.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Day 1 to Day 211
Population: Safety Analysis Set (SAS): Included all participants randomized in Phase 2b or 3 who received at least one dose of CVnCoV or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 19787 | 19753
Participants
  Any Medically-attended AE | 2555 | 2084
  Any Related Medically-attended AE | 505 | 138

3. Primary Outcome: Number of Participants Who Experienced One or More Serious AE (SAE)
Description: An SAE was defined as any untoward medical occurrence that, at any dose:
  * Resulted in death.
  * Was life-threatening.
  * Required inpatient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent disability/incapacity.
  * Was a congenital anomaly/birth defect in the offspring of the participant.
  * Was an important medical event.
  The Investigator assessed the relationship between trial vaccine and occurrence of each SAE.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Day 1 to Day 393
Population: SAS: Included all participants randomized in Phase 2b or 3 who received at least one dose of CVnCoV or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 19787 | 19753
Participants
  Any SAE | 149 | 111
  Any Related SAE | 8 | 1

4. Primary Outcome: Intensity of SAEs as Per Investigator Assessment
Description: An SAE was defined as any untoward medical occurrence that, at any dose:
  * Resulted in death.
  * Was life-threatening.
  * Required inpatient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent disability/incapacity.
  * Was a congenital anomaly/birth defect in the offspring of the participant.
  * Was an important medical event.
  The Investigator made an assessment of intensity of each SAE reported during the trial. Each SAE was graded from Mild (Grade 1) to Severe (Grade 3), where higher grades indicated a worse outcome.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Day 1 to Day 393
Population: SAS: Included all participants randomized in Phase 2b or 3 who received at least one dose of CVnCoV or placebo. Only participants who experienced SAEs were included.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 149 | 111
Participants
  Mild (Grade 1) | 21 | 10
  Moderate (Grade 2) | 50 | 35
  Severe (Grade 3) | 74 | 66
  Missing | 4 | 0

5. Primary Outcome: Number of Participants Who Experienced One or More Adverse Event of Special Interest (AESI)
Description: AESIs included:
  * AEs with a suspected immune-medicated etiology.
  * Other AEs relevant to SARS-CoV-2 vaccine development or the target disease.
  The Investigator assessed the relationship between trial vaccine and occurrence of each AESI.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Day 1 to Day 393
Population: SAS: Included all participants randomized in Phase 2b or 3 who received at least one dose of CVnCoV or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 19787 | 19753
Participants
  Any AESI | 64 | 47
  Any Related AESI | 19 | 5

6. Primary Outcome: Number of Participants Who Experienced a Fatal SAE
Description: A fatal SAE was defined as an SAE that resulted in death.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Day 1 to Day 393
Population: SAS: Included all participants randomized in Phase 2b or 3 who received at least one dose of CVnCoV or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 19787 | 19753
Participants | 11 | 12

7. Primary Outcome: Phase 2b Participants Only: Number of Participants Who Experienced One or More Solicited AE
Description: Solicited local AEs (injection site pain, redness, swelling, and itching) and solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) were recorded on the day of vaccination and the following 7 days using an eDiary.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Up to 7 days after vaccination (Days 1 to 7 and Days 29 to 36)
Population: The SASsol: Included all phase 2b participants of the SAS with at least one diary collection indicating the occurrence or lack of occurrence of solicited AEs.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 2003 | 1978
Participants
  Any Solicited Local AE | 1699 | 477
  Any Solicited Systemic AE | 1881 | 1255

8. Primary Outcome: Phase 2b Participants Only: Intensity of Solicited AEs as Per Investigator Assessment
Description: Solicited local AEs (injection site pain, redness, swelling, and itching) and solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) were recorded on the day of vaccination and the following 7 days using an eDiary.
  The Investigator made an assessment of intensity of each solicited AE reported during the trial. Each solicited AE was graded from Mild (Grade 1) to Severe (Grade 3), where higher grades indicated a worse outcome.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Up to 7 days after vaccination (Days 1 to 7 and Days 29 to 36)
Population: The SASsol: Included all phase 2b participants of the SAS with at least one diary collection indicating the occurrence or lack of occurrence of solicited AEs. Only participants who experienced solicited AEs were included.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 1933 | 1344
Participants
  Any Solicited Local AEs: number analyzed (Participants) | 1699 | 477
  Any Solicited Local AEs: Mild (Grade 1) | 1226 | 452
  Any Solicited Local AEs: Moderate (Grade 2) | 448 | 24
  Any Solicited Local AEs: Severe (Grade 3) | 25 | 1
  Any Solicited Systemic AEs: number analyzed (Participants) | 1881 | 1255
  Any Solicited Systemic AEs: Mild (Grade 1) | 376 | 708
  Any Solicited Systemic AEs: Moderate (Grade 2) | 969 | 487
  Any Solicited Systemic AEs: Severe (Grade 3) | 536 | 60

9. Primary Outcome: Phase 2b Participants Only: Duration of Solicited AEs
Description: Solicited local AEs (injection site pain, redness, swelling, and itching) and solicited systemic AEs (fever, headache, fatigue, chills, myalgia, arthralgia, nausea/vomiting, and diarrhea) were recorded on the day of vaccination and the following 7 days using an eDiary. Duration is calculated as consecutive days with a respective solicited AE regardless of the grade of the AE. AEs ongoing after Day 8 are included. In each case only the longest consecutive duration is displayed.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Up to 7 days after vaccination (Days 1 to 7 and Days 29 to 36)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 1933 | 1344
days
  Solicited Local AEs - Injection Site Pain: number analyzed (Participants) | 1674 | 417
  Solicited Local AEs - Injection Site Pain | 2.3 (1.24) | 1.5 (1.24)
  Solicited Local AEs - Redness: number analyzed (Participants) | 89 | 25
  Solicited Local AEs - Redness | 2.2 (2.32) | 2.1 (1.99)
  Solicited Local AEs - Swelling: number analyzed (Participants) | 149 | 17
  Solicited Local AEs - Swelling | 1.7 (0.97) | 1.2 (0.56)
  Solicited Local AEs - Itching: number analyzed (Participants) | 141 | 93
  Solicited Local AEs - Itching | 1.6 (1.20) | 1.4 (1.42)
  Solicited Systemic AEs - Fever: number analyzed (Participants) | 617 | 13
  Solicited Systemic AEs - Fever | 1.3 (0.52) | 1.0 (0.00)
  Solicited Systemic AEs - Headache: number analyzed (Participants) | 1541 | 806
  Solicited Systemic AEs - Headache | 2.0 (1.41) | 1.8 (2.45)
  Solicited Systemic AEs - Fatigue: number analyzed (Participants) | 1603 | 845
  Solicited Systemic AEs - Fatigue | 2.3 (2.84) | 2.0 (2.25)
  Solicited Systemic AEs - Chills: number analyzed (Participants) | 1011 | 162
  Solicited Systemic AEs - Chills | 1.3 (0.67) | 1.4 (0.83)
  Solicited Systemic AEs - Myalgia: number analyzed (Participants) | 1327 | 378
  Solicited Systemic AEs - Myalgia | 1.8 (1.08) | 1.6 (1.13)
  Solicited Systemic AEs - Arthralgia: number analyzed (Participants) | 578 | 148
  Solicited Systemic AEs - Arthralgia | 1.6 (0.98) | 1.6 (1.19)
  Solicited Systemic AEs - Nausea/Vomiting: number analyzed (Participants) | 414 | 151
  Solicited Systemic AEs - Nausea/Vomiting | 1.5 (0.97) | 1.3 (0.82)
  Solicited Systemic AEs - Diarrhea: number analyzed (Participants) | 376 | 224
  Solicited Systemic AEs - Diarrhea | 1.4 (0.95) | 1.3 (0.90)

10. Primary Outcome: Phase 2b Participants Only: Number of Participants Who Experienced One or More Unsolicited AE
Description: eDiaries were used for collection of unsolicited AEs on each vaccination day and the following 28 days. In addition, participants received a prompt (by e.g., a phone call or text message) to verify whether the participants had any health concerns since the last visit. The Investigator assessed the relationship between trial vaccine and each occurrence of each AE.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Up to 28 days after vaccination (Days 1 to 29 and Days 29 to 57)
Population: SAS 2: Included all Phase 2b participants of the SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 2007 | 1987
Participants
  Any Unsolicited AE | 1016 | 911
  Any Related Unsolicited AE | 511 | 269

11. Primary Outcome: Phase 2b Participants Only: Intensity of Unsolicited AEs as Per Investigator Assessment
Description: eDiaries were used for collection of unsolicited AEs on each vaccination day and the following 28 days. In addition, participants received a prompt (by e.g., a phone call or text message) to verify whether the participants had any health concerns since the last visit.
  The Investigator made an assessment of intensity of each unsolicited AE reported during the trial. Each unsolicited AE was graded from Mild (Grade 1) to Severe (Grade 3), where higher grades indicated a worse outcome.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Up to 28 days after vaccination (Days 1 to 29 and Days 29 to 57)
Population: SAS 2: Included all Phase 2b participants of the SAS.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 1016 | 911
Participants
  Mild (Grade 1) | 712 | 641
  Moderate (Grade 2) | 259 | 225
  Severe (Grade 3) | 44 | 38
  Missing | 1 | 7

12. Primary Outcome: Number of Participants Who Experienced One or More AEs Leading to Vaccine Withdrawal or Trial Discontinuation
Description: Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Day 1 to Day 393
Population: SAS: Included all participants randomized in Phase 2b or 3 who received at least one dose of CVnCoV or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 19787 | 19753
Participants
  Any AE Leading to Vaccine Withdrawal | 32 | 33
  Any AE Leading to Withdrawal From Trial | 17 | 16

13. Secondary Outcome: Number of Participants Who Experienced a First Episode of Virologically-confirmed (RT-PCR Positive) Moderate to Severe Case of COVID-19
Description: Moderate cases defined by any 1 of the following:
  * Shortness of breath/difficulty breathing
  * Respiratory rate ≥20 to <30 breaths per min
  * Abnormal SpO2 but still >93% on room air at sea level
  * Clinical/radiographic evidence of lower respiratory tract disease
  * Radiologic evidence of DVT
  Severe cases defined by any 1 of the following:
  * Clinical signs at rest indicative of severe systemic illness (respiratory rate ≥ 30breaths per minute, heart rate ≥125 per minute, SpO2 ≤93% on room air at sea level or PaO2/FIO2 <300 mm Hg)
  * Respiratory failure (defined as needing high flow-oxygen, noninvasive ventilation, mechanical ventilation or ECMO)
  * Evidence of shock (SBP <90mm Hg, DBP <60 mmHg or requiring vasopressors)
  * Significant renal, hepatic, or neurologic dysfunction
  * Admission to ICU
  * Death
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Day 44 to Day 393
Population: EAS: All participants randomized in Phase 2b or Phase 3 who received both doses of trial vaccine, had not developed a virologically-confirmed case of COVID-19 before trial entry or before 15 days after the second vaccination, & were SARS-CoV-2 naïve at baseline and Day 43. Participants must have not developed an asymptomatic case of SARS-CoV-2, not stopped the trial, not received an AV for preventing COVID-19 or not been unblinded prior to 15 days after the second vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 12851 | 12211
Participants | 12 | 37
Statistical Analysis 1: Comparison: CVnCoV 12 μg Vaccine vs Placebo; Proportion of cases coming from the CVnCoV group among all cases; Test type: Superiority; Proportion = 0.245, 95% CI 2-sided [0.133 to 0.389] — Derived from an exact 2-sided 95% Pearson-Clopper CI on proportion of cases coming from the CVnCoV group among all cases
Statistical Analysis 2: Comparison: CVnCoV 12 μg Vaccine vs Placebo; VE calculated as VE = 1 - p/(1-p) *1/r where p represents the proportion of cases coming from the CVnCoV group among all cases and r represents the ratio of total follow-up time of subjects in the CVnCoV group over the total follow-up time of subjects in the placebo group; Test type: Superiority; Vaccine Efficacy = 70.7, 95% CI 2-sided [42.5 to 86.1] — 2-sided 95% CI on VE, derived from the exact 2-sided 95% Pearson-Clopper CI on proportion of cases coming from the CVnCoV group among all cases

14. Secondary Outcome: Number of Participants Who Experienced a First Episode of Virologically-confirmed (RT-PCR Positive) Severe Case of COVID-19
Description: Severe COVID-19 cases were defined by any one of the following:
  * Clinical signs at rest indicative of severe systemic illness (respiratory rate ≥ 30 breaths per minute, heart rate ≥ 125 per minute, SpO2 ≤ 93% on room air at sea level or PaO2/FIO2 < 300 mm Hg).
  * Respiratory failure (defined as needing high flow-oxygen, noninvasive ventilation, mechanical ventilation or ECMO).
  * Evidence of shock (SBP < 90mm Hg, DBP < 60 mmHg, or requiring vasopressors).
  * Significant renal, hepatic, or neurologic dysfunction
  * Admission to intensive care unit (ICU).
  * Death.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Day 44 to Day 393
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 12851 | 12211
Participants | 4 | 10
Statistical Analysis 1: Comparison: CVnCoV 12 μg Vaccine vs Placebo; Proportion of cases coming from the CVnCoV group among all cases; Test type: Superiority; Proportion = 0.286, 95% CI 2-sided [0.084 to 0.581] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: CVnCoV 12 μg Vaccine vs Placebo; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; Vaccine Efficacy = 63.8, 95% CI 2-sided [-25.5 to 91.7] — [estimate comment as in outcome 13, analysis 2]

15. Secondary Outcome: Number of Participants Who Experienced a First Episode of Virologically-confirmed (RT-PCR Positive) Case of COVID-19 of Any Severity Due to Infection With "Wild Type" and "Alpha" SARS-CoV-2 Strains in SARS-CoV-2 Naïve Participants
Description: The characterization of SARS-CoV-2 variants were implemented by viral whole genome sequencing of nasopharyngeal swab samples of participants followed by comparison with previously sequenced and typified genomes. The following phylogenetic clustering was applied:
  1. "Wild type" virus: WT/D614G, lineages A.1/B.1 without the variant of concerns (VOCs) (i.e., without B.1.1.7 [Alpha], B.1.351 [Beta], B.1.429 [Epsilon]).
  2. "UK" VOC: B.1.1.7 (Alpha).
  A case of COVID-19 was defined as follows:
  * Virologically-confirmed case of COVID-19 defined as a positive SARS-CoV-2 specific RT-PCR test in a person with clinically symptomatic COVID-19.
  * Symptom onset ≥ 15 days after second vaccination.
  * First episode of virologically-confirmed COVID-19.
  * Participant was SARS-CoV-2 naïve at baseline and Day 43.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Day 44 to Day 393
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 12851 | 12211
Participants | 29 | 56
Statistical Analysis 1: Comparison: CVnCoV 12 μg Vaccine vs Placebo; Proportion of cases coming from the CVnCoV group among all cases; Test type: Superiority; Proportion = 0.341, 95% CI 2-sided [0.242 to 0.452] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: CVnCoV 12 μg Vaccine vs Placebo; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; Vaccine Efficacy = 53.2, 95% CI 2-sided [25.4 to 71.2] — [estimate comment as in outcome 13, analysis 2]

16. Secondary Outcome: Number of Participants Aged ≥ 61 Who Experienced a First Episode of Virologically-confirmed (RT-PCR Positive) Case of COVID-19 of Any Severity
Description: A case of COVID-19 was defined as follows:
  * Virologically-confirmed case of COVID-19 (of any severity) defined as a positive SARS-CoV-2 specific RT-PCR test in a person with clinically symptomatic COVID-19.
  * Symptom onset ≥ 15 days after second trial vaccination.
  * First episode of virologically-confirmed COVID-19, i.e. the participant must not have had a history of virologically-confirmed COVID-19 illness at enrollment or have had developed a case of virologically-confirmed COVID-19 before 15 days after the second trial vaccination.
  * Participant was SARS-CoV-2 naïve at baseline and Day 43 (defined as seronegative to N protein in the blood samples collected at baseline and Day 43).
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Day 44 to Day 393
Population: The EAS including only participants who were aged ≥ 61.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 1319 | 1180
Participants | 12 | 9
Statistical Analysis 1: Comparison: CVnCoV 12 μg Vaccine vs Placebo; Proportion of cases coming from the CVnCoV group among all cases; Test type: Superiority; Proportion = 0.571, 95% CI 2-sided [0.340 to 0.782] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: CVnCoV 12 μg Vaccine vs Placebo; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; Vaccine Efficacy = -11.8, 95% CI 2-sided [-200.5 to 56.7] — [estimate comment as in outcome 13, analysis 2]

17. Secondary Outcome: Burden of Disease (BoD) Score #1 Based on First Episodes of Virologically-confirmed (RT-PCR Positive) Cases of COVID-19
Description: Score #1 was defined as no disease (not infected or asymptomatic infection) = 0; mild or moderate disease = 1; severe disease = 2.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Day 44 to Day 393
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 12851 | 12211
Participants
  0 | 12768 | 12066
  1 | 79 | 135
  2 | 4 | 10

18. Secondary Outcome: BoD Score #2 Based on First Episodes of Virologically-confirmed (RT-PCR Positive) Cases of COVID-19
Description: Score #2 was defined as no disease (not infected or asymptomatic infection) = 0; disease without hospitalization = 1; disease with hospitalization = 2; death = 3.
  Participants were censored at the first day after unblinding or at the day after receiving the authorized/licensed vaccine, whichever was earlier.
Time Frame: Day 44 to Day 393
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 12851 | 12211
Participants
  0 | 12768 | 12066
  1 | 82 | 143
  2 | 0 | 2
  3 | 1 | 0

19. Secondary Outcome: SARS-CoV-2 Receptor Binding Domain (RBD) of Spike (S) Protein Antibody Levels on Days 1, 29, 43, 120 and 211
Description: Titers of IgG antibodies directed against the SARS-CoV-2 RBD of Spike Protein antigen were measured by enzyme- linked immunosorbent assay (ELISA) and expressed as geometric mean of titers (GMT) with 95% confidence interval (CI), by group. Individual values below the lower limit of quantification (LLOQ) were set to half of the LLOQ. Only participants seronegative at baseline with evaluable samples at each visit are included. Participants who tested positive for SARS-CoV-2 via PCR or N-protein antibodies had their data included up to the point of positive test result or symptom onset.
  Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Days 1 (baseline), 29, 43, 120 and 211
Population: Per Protocol Immunogenicity (PPI) Set: Included all Phase 2b participants from the Immunogenicity Subset who received both doses as randomized and within the specified windows, had no important protocol deviations that impacted immunogenicity outcomes, did not receive medical treatments that interfered with the proposed immunogenicity measurements and had at least one blood sample collected at baseline and starting at 14 days post-second vaccination available for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 544 | 525
titers
  Day 1 | 50.791 [50.151 to 51.439] | 50.763 [50.079 to 51.456]
  Day 29: number analyzed (Participants) | 536 | 516
  Day 29 | 54.090 [52.213 to 56.034] | 50.734 [50.074 to 51.403]
  Day 43: number analyzed (Participants) | 518 | 498
  Day 43 | 734.657 [645.552 to 836.061] | 50.902 [50.082 to 51.737]
  Day 120: number analyzed (Participants) | 432 | 245
  Day 120 | 227.439 [203.647 to 254.011] | 57.357 [52.843 to 62.257]
  Day 211: number analyzed (Participants) | 27 | 7
  Day 211 | 371.341 [161.098 to 855.966] | 107.556 [23.919 to 483.648]

20. Secondary Outcome: Percentage of Participants Seroconverting to SARS-CoV-2 RBD of S Protein Antibodies on Days 29, 43, 120 and 211
Description: Titers of IgG antibodies directed against the SARS-CoV-2 RBD of Spike Protein antigen were measured by ELISA. Percentage with 95% CI of participants for whom a seroconversion was observed is presented by group. In participants who tested seronegative to the N protein for SARS-CoV-2 at baseline, seroconversion was defined as a fold increase above 1 in antibody titer against SARS-CoV-2 RBD of S protein. Only participants seronegative at baseline with evaluable samples at each visit are included. Participants who tested positive for SARS-CoV-2 via PCR or N-protein antibodies had their data included up to the point of positive test result or symptom onset. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Baseline and Days 29, 43, 120 and 211
Population: PPI Set: Included all Phase 2b participants seronegative at baseline from the Immunogenicity Subset who received both doses as randomized & within the specified windows, had no important protocol deviations that impacted immunogenicity outcomes, did not receive medical treatments that interfered with the proposed immunogenicity measurements and had at least one blood sample collected at baseline and starting at 14 days post-second vaccination available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 536 | 516
percentage of participants
  Day 29 | 4.3 [2.7 to 6.4] | 0.4 [0.0 to 1.4]
  Day 43: number analyzed (Participants) | 518 | 498
  Day 43 | 87.1 [83.9 to 89.8] | 0.6 [0.1 to 1.8]
  Day 120: number analyzed (Participants) | 432 | 245
  Day 120 | 72.2 [67.7 to 76.4] | 4.9 [2.6 to 8.4]
  Day 211: number analyzed (Participants) | 27 | 7
  Day 211 | 66.7 [46.0 to 83.5] | 28.6 [3.7 to 71.0]

21. Secondary Outcome: SARS-CoV-2 Viral Neutralizing Antibody Levels on Days 1, 29, 43, 120 and 211
Description: Titers of viral neutralizing antibodies were determined by an activity assay and expressed as GMT with 95% CI, by group. Individual values below the LLOQ were set to half of the LLOQ. Only participants seronegative at baseline with evaluable samples at each visit are included. Participants who have tested positive for SARS-CoV-2 via PCR or N-protein antibodies have their data included up to the point of positive test result or symptom onset. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Days 1 (baseline), 29, 43, 120 and 211
Population: PPI Set: Included all Phase 2b participants from the Immunogenicity Subset who received both doses as randomized and within the specified windows, had no important protocol deviations that impacted immunogenicity outcomes, did not receive medical treatments that interfered with the proposed immunogenicity measurements and had at least one blood sample collected at baseline and starting at 14 days post-second vaccination available for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 544 | 525
titers
  Day 1 (Baseline) | 5.016 [4.993 to 5.039] | 5.007 [4.994 to 5.020]
  Day 29: number analyzed (Participants) | 536 | 516
  Day 29 | 5.141 [5.022 to 5.263] | 5.030 [4.995 to 5.066]
  Day 43: number analyzed (Participants) | 518 | 498
  Day 43 | 18.211 [16.394 to 20.230] | 5.049 [5.003 to 5.096]
  Day 120: number analyzed (Participants) | 432 | 245
  Day 120 | 7.105 [6.640 to 7.603] | 5.136 [5.008 to 5.267]
  Day 211: number analyzed (Participants) | 27 | 7
  Day 211 | 14.325 [7.183 to 28.565] | 6.729 [4.209 to 10.757]

22. Secondary Outcome: Percentage of Participants Seroconverting to SARS-CoV-2 Viral Neutralizing Antibodies on Days 29, 43, 120 and 211
Description: Titers of viral neutralizing antibodies were determined by an activity assay. Percentage with 95% CI of participants for whom a seroconversion was observed is presented by group. In participants who tested seronegative to the N protein for SARS-CoV-2 at baseline, seroconversion was defined as a fold increase above 1 in antibody titer against SARS-CoV-2 neutralizing antibody titer. Only participants seronegative at baseline with evaluable samples at each visit are included. Participants who have tested positive for SARS-CoV-2 via PCR or N-protein antibodies have their data included up to the point of positive test result or symptom onset. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Baseline and Days 29, 43, 120 and 211
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
Number analyzed (Participants) | 536 | 516
percentage of participants
  Day 29 | 1.5 [0.6 to 2.9] | 0.6 [0.1 to 1.7]
  Day 43: number analyzed (Participants) | 518 | 498
  Day 43 | 65.1 [60.8 to 69.2] | 1.0 [0.3 to 2.3]
  Day 120: number analyzed (Participants) | 432 | 245
  Day 120 | 24.8 [20.8 to 29.1] | 2.0 [0.7 to 4.7]
  Day 211: number analyzed (Participants) | 27 | 7
  Day 211 | 33.3 [16.5 to 54.0] | 28.6 [3.7 to 71.0]

ADVERSE EVENTS:
Time Frame: Day 1 to Day 393
Description: Participants who became unblinded and/or received a licensed/authorized vaccine were censored at the day after unblinding or at the day after receiving the licensed/authorized vaccine, whichever is earlier. All-cause mortality includes non-censored data.
Arm/Group | CVnCoV 12 μg Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 17/19787 | 14/19753
Serious Adverse Events (participants affected / at risk) | 149/19787 | 111/19753
Other Adverse Events (participants affected / at risk) | 3144/19787 | 1853/19753
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CVnCoV 12 μg Vaccine (N=19787) | Placebo (N=19753)
Appendicitis (Infections and infestations) | 8 | 3
COVID-19 pneumonia (Infections and infestations) | 5 | 4
COVID-19 (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 1
Complicated appendicitis (Infections and infestations) | 2 | 0
Hantaviral infection (Infections and infestations) | 2 | 0
Liver abscess (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 2
Abscess (Infections and infestations) | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Bartholin's abscess (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Haemorrhagic fever with renal syndrome (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 1 | 0
Oophoritis (Infections and infestations) | 1 | 0
Pelvic infection (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Q fever (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Salpingitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 2 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 2
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1
Laryngeal injury (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ovarian germ cell teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neurofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Retroperitoneal neoplasm metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 4
Pregnancy with injectable contraceptive (Pregnancy, puerperium and perinatal conditions) | 2 | 3
Pregnancy on oral contraceptive (Pregnancy, puerperium and perinatal conditions) | 4 | 0
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 | 2
Abortion (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Silent myocardial infarction (Cardiac disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 2
Carotid sinus syndrome (Nervous system disorders) | 1 | 0
Cerebral ventricle dilatation (Nervous system disorders) | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Complex regional pain syndrome (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Multifocal motor neuropathy (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 1
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 1 | 0
Peripheral nerve paresis (Nervous system disorders) | 1 | 0
Radial nerve palsy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Status migrainosus (Nervous system disorders) | 0 | 1
Thalamic infarction (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1
Colitis microscopic (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0
Malocclusion (Gastrointestinal disorders) | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 3
Cholecystitis acute (Hepatobiliary disorders) | 4 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary cyst (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Plica syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 4
Calculus urinary (Renal and urinary disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
IgA nephropathy (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 3
Suicide attempt (Psychiatric disorders) | 1 | 2
Suicidal ideation (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 | 0
Self-injurious ideation (Psychiatric disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 2 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Fallopian tube cyst (Reproductive system and breast disorders) | 1 | 0
Hydrosalpinx (Reproductive system and breast disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 2 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Optic nerve disorder (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Basedow's disease (Endocrine disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
HIV test positive (Investigations) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVnCoV 12 μg Vaccine (N=19787) | Placebo (N=19753)
Chills (General disorders) | 1439 (2065) | 240 (286)
Fatigue (General disorders) | 1893 (3200) | 1019 (1483)
Injection site pain (General disorders) | 2008 (3231) | 537 (644)
Pyrexia (General disorders) | 1305 (1700) | 95 (102)
Myalgia (Musculoskeletal and connective tissue disorders) | 1728 (2588) | 509 (634)
Headache (Nervous system disorders) | 2310 (3911) | 1225 (1805)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT04652102/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT04652102/SAP_001.pdf